CLINICAL TRIAL: NCT00925041
Title: Clinical Evaluation of the Vedera KXS for the Treatment of Spherical Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avedro T1
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kxl Vedera (Experimental)
  Interventions: Device: Vedera KXS

INTERVENTIONS:
Device: Vedera KXS — one treatment with the Vedera KXS

SUMMARY:
The objective of this clinical investigation is to evaluate the safety and efficacy of the Vedera KXS in sighted eyes for the correction of spherical myopia.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing surgery for the correction of myopia
* Intended treatment from -0.5 to -6.0 D of spherical myopia
* Must have 0.50 D or less astigmatic component.
* Must have bilateral physiologic myopia
* BSCVA of 20/25 or better in each eye
* Must have had a stable refraction (0.5 D or less change in spheroequivalent) for at least one year, objectively documented (by previous clinical records, eyeglass prescriptions, etc. over one year old)
* Patients who are contact lens wearers must have hard or gas permeable lenses discontinued for two weeks and soft lenses discontinued for three days prior to the preoperative evaluation
* Must be at least 18 years of age
* Corneal topography must be normal, as judged by the investigator
* Must have a minimal corneal thickness of 475 microns
* Must sign a written Informed Consent form acknowledging their awareness of their participation in this study, the alternative treatments available, the risks involved, and the investigative nature of the procedure, and other issues which conform to the standard of care for Informed Consent practices
* Must be willing and capable of returning for scheduled follow-up examinations for 24 months after treatment

Exclusion Criteria:

* Patients who are unable or unwilling to sign the informed consent form.
* Anterior segment pathology
* Residual, recurrent or active ocular disease
* Patients who have undergone previous intraocular or corneal surgery involving the stroma in the eye to be operated.
* History of herpes keratitis
* Patients with diagnosed autoimmune disease, systemic connective tissue diseases or atopic syndrome, diabetes mellitus, or taking systemic medications (i.e., corticosteroids or antimetabolites) likely to affect wound healing.
* Irregular central keratometry/topography readings with irregular topography patterns or keratometry mires, including signs of keratoconus.
* Patients with known sensitivity to study medications.
* Intraocular pressure of > 23 mm Hg by Goldmann applanation tonometry, a history of glaucoma, or glaucoma suspect.
* Women who are pregnant or nursing or who plan to become pregnant over the course of their participation in this investigation.
* Participation in other ophthalmic clinical trials during this clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
UCVA 20/40 or better | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beyoglu Eye Research and Education Hospital, Istanbul, Turkey (Türkiye)